CLINICAL TRIAL: NCT07322354
Title: A Pragmatic Randomized Controlled Trial on the Effectiveness of a Multi-Modal Rest Cabin in Boosting Worker Well-Being
Brief Title: Effectiveness of a Multi-Modal Workplace Rest Cabin on Worker Well-Being
Acronym: RECHARJME-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Simon Coulombe, Full Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Recharjme-RCT-2024; 2023-2766 (Other: Comité d'éthique de la santé des populations et première ligne (CIUSSS-CN))
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Employee Well-being; Work-related Outcomes
Keywords: Workplace well-being; Rest cabin; Micro-breaks; Burnout; Workplace intervention; Recovery at work; Employee mental health; Mindful attention awareness; Psychological detachment from work
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest Cabin Use (Experimental): Participants are encouraged to use the Recharjme cabin for one month (four weeks) at a frequency of three times a week, preferably between 9 a.m. and 4 p.m.
  Interventions: Device: Recharjme Multi-Modal Rest Cabin
- Waiting List Control (No Intervention): No cabin access for four weeks.

INTERVENTIONS:
Device: Recharjme Multi-Modal Rest Cabin — Enclosed workplace cabin with guided meditation, massage, luminotherapy, and zero-gravity chair.
  Arms: Rest Cabin Use

SUMMARY:
This study examines whether access to a rest cabin in the workplace supports employee well-being. Employees of a Canadian insurance company are randomly assigned to one of two groups: immediate access to the rest cabin or a waiting-list control group that receives access after one month. The rest cabin is installed directly in the workplace and can be reserved for short sessions during the workday. It offers multiple relaxation options, including guided meditation, massage therapy, light therapy, and a zero-gravity chair. Employees choose which options to use during each session. Participants complete questionnaires before group assignment and again one month later. Employees who receive immediate access to the cabin also complete additional follow-up questionnaires at later time points. The study compares changes in general well-being and work-related outcomes between employees who have access to the cabin and those who do not during the initial study period.

DETAILED DESCRIPTION:
This pragmatic randomized controlled trial evaluates the effects of a multi-modal rest cabin on general and work-related well-being among employees of a Canadian insurance company. The study takes place in real-world workplace settings across multiple office locations. After providing informed consent, participants complete a baseline survey assessing general well-being and work-related outcomes. Participants are then randomly assigned to one of two conditions: (1) immediate access to the rest cabin or (2) a waiting-list control condition with delayed access. Employees assigned to the immediate-access group are encouraged to use the rest cabin over a four-week period. Cabin sessions are self-scheduled during work hours and are designed to be brief. The rest cabin is fully enclosed and located within the workplace. It includes several relaxation modalities, such as guided meditation, massage therapy, light therapy, and a zero-gravity chair. Participants are free to select and combine modalities based on their preferences during each session. Participants in both the immediate-access group and the waiting-list control group complete a follow-up survey one month after the baseline assessment. To examine whether any observed changes are maintained over time, participants in the immediate-access group also complete additional follow-up surveys two months and four months after baseline. It is hypothesized that workers in the experimental (vs. control) group would have better changes in scores in their general (positive and negative affect, flourishing, anxiety, depression, mindful attention awareness, insomnia) and workplace (thriving at work, burnout, absenteeism, presenteeism, job satisfaction, psychological detachment from work) positive and negative well-being when comparing Time 1 (follow-up survey) to Time 0 (baseline) (H1). Specific to those in the experimental condition, it is hypothesized that: positive changes observed following cabin use (at Time 1) would remain evident at the subsequent follow-up timepoints (Times 2 and 3), relative to baseline (H2), and changes in well-being outcomes between Time 1 and Time 0 would be greater for those who have used the cabin more often (H3). It is also hypothesized that: 4) the change in outcomes between T1 and T0 associated with being in the experimental (vs. control) condition (as discussed in H1) would be mediated by changes in psychological detachment from work and mindfulness awareness (H4), and 5) the relationship between cabin use frequency and changes in well-being outcomes (as discussed in H3) would be mediated by changes in psychological detachment and mindfulness awareness (also between T1 and T0; H5).

ELIGIBILITY:
Inclusion Criteria:

* Employee of participating insurance company
* Aged 18 or older

Exclusion Criteria:

* Mental health leave in past year
* Diagnosed mental health disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Presenteeism (impaired productivity and troublesome symptoms at work) | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the Employment Absence and Productivity Scale; Min.: 1; Max.: 5; Higher scores indicating a more negative outcome.
Absenteeism | Time 0 (baseline) to time 3 (four months after baseline)
  Calculation based on the World Health Organization Health and Work Performance Questionnaire; Min.: 0; Max.: 100; Higher scores indicating a more negative outcome.
Job satisfaction | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using an adapted item from Life in Transition Survey; Min.: 1; Max.: 5; Higher scores indicating a more positive outcome.
Anxiety and depression | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the two subscales of the Patient Health Questionnaire-4; Min.: 1; Max.: 4; Higher scores indicating a more negative outcome.
Insomnia | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the Insomnia Severity Index; Min.: 0; Max.: 4; Higher scores indicating a more negative outcome.
Burnout (physical fatigue, cognitive weariness, emotional exhaustion) | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the three subscales of the Shirom-Melamed Burnout Measure; Min.: 1; Max.: 7; Higher scores indicating a more negative outcome.
Flourishing | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the Flourishing Scale; Min.: 1; Max.: 7; Higher scores indicating a more positive outcome.
Thriving at work | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using Index of Psychological Well-Being at Work (Thriving at Work Subscale); Min.: 0; Max.: 5; Higher scores indicating a more positive outcome.
Mindful attention awareness | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the Mindful Attention Awareness Scale (Carlson & Brown, 2005); Min.: 1; Max.: 6; Higher scores indicating a more positive outcome.
Psychological detachment from work | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using adapted items from Recovery Experience Questionnaire; Min.: 1; Max.: 5; Higher scores indicating a more positive outcome.
Positive and Negative Affect | Time 0 (baseline) to time 3 (four months after baseline)
  Measured using the two subscales of the Positive and Negative Affect Schedule; Min.: 1; Max.: 5; For positive affect: higher scores indicating a more positive outcome; For negative affect, higher scores indicating a more negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Coulombe, PhD, Principal Investigator — Laval University
Locations (4):
- Canada (4):
  - Worksite 3, Mississauga, Ontario
  - Worksite 3, Longueuil, Quebec
  - Worksite 1, Québec, Quebec
  - Worksite 2, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ipsos. (n.d.). Life in transition survey IV for the European Bank for Reconstruction and Development: Technical report. The European Bank for Reconstruction and Development. https://www.ebrd.com/content/dam/ebrd_dxp/assets/pdfs/office-of-the-chief-economist/publications/life-in-transition-survey-iv/LITS-IV-Technical-report.pdf
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Sonnentag S, Fritz C. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. J Occup Health Psychol. 2007 Jul;12(3):204-21. doi: 10.1037/1076-8998.12.3.204. PMID 17638488
- [Background] Carlson LE, Brown KW. Validation of the Mindful Attention Awareness Scale in a cancer population. J Psychosom Res. 2005 Jan;58(1):29-33. doi: 10.1016/j.jpsychores.2004.04.366. PMID 15771867
- [Background] Dagenais-Desmarais, V., & Savoie, A. (2012). What is psychological well-being, really? A grassroots approach from the organizational sciences. Journal of Happiness Studies, 13(4), 659-684.
- [Background] Shirom, A., & Melamed, S. (2006). A comparison of the construct validity of two burnout measures in two groups of professionals. International Journal of Stress Management, 13(2), 176-200
- [Background] Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi, D. W., Oishi, S., & Biswas-Diener, R. (2010). New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social Indicators Research, 97(2), 143-156.
- [Background] Sassi, N., & Neveu, J. P. (2010). Traduction et validation d'une nouvelle mesure d'épuisement professionnel: Le shirom-melamed burnout measure. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 42(3), 177-184.
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] Lam RW, Michalak EE, Yatham LN. A new clinical rating scale for work absence and productivity: validation in patients with major depressive disorder. BMC Psychiatry. 2009 Dec 3;9:78. doi: 10.1186/1471-244X-9-78. PMID 19958540